CLINICAL TRIAL: NCT03788343
Title: PICO: Phenylalanine and Its Impact on Cognition - Impact of Phenylalanine on Cognitive, Cerebral and Neurometabolic Parameters in Adult Patients With Phenylketonuria
Brief Title: Phenylalanine and Its Impact on Cognition
Acronym: PICO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018-01609; 3837 (Other: Inselspital, Bern University Hospital)
Record Dates: First submitted 2018-12-17; First posted 2018-12-27 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Phenylketonuria
Keywords: Phenylketonuria; PKU; Phenylalanine; Diet; Neuropsychology; Working Memory; Neuroimaging
MeSH Terms: conditions — Phenylketonurias | interventions — Phenylalanine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenylalanine (Experimental): Capsules containing 250 mg Phenylalanine (Phe). The daily dose will be chosen according to gender and weight at the time of T1 and will be divided in 3 separate doses. The assigned dose of the IMP will be kept throughout the whole study and weight fluctuations will not be considered.
  Female
  <60 kg: 1500 mg per day (divided in 3 doses): 250 mg 2-2-2-0
  ≥60 kg: 2000 mg per day (divided in 3 doses): 250 mg 2-2-4-0
  Male
  <60 kg: 2500 mg per day (divided in 3 doses): 250 mg 4-2-4-0
  ≥60 kg: 3000 mg per day (divided in 3 doses): 250 mg 4-4-4-0
  Phe capsules can be ingested before, during or after a meal or together with other amino acid supplements. The last capsule of the given intervention period will be timed to be ingested with the last meal before the study visit.
  Patients will take Phe for 4 weeks.
  Interventions: Dietary Supplement: Phenylalanine
- Placebo (Placebo Comparator): Capsules containing 250mg Placebo. Placebo capsules will be administered in identical manner to Phe capsules.
  Patients will take the Placebo for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Phenylalanine — The study product Phenylalanine, a dietary supplement, is authorized in Switzerland, but not designated for this patient group.
  Arms: Phenylalanine
Drug: Placebo — Placebo capsules are indistinguishable in their appearance from Phe capsules
  Arms: Placebo

SUMMARY:
The PICO-Study is a randomized, placebo-controlled, crossover, non-inferiority trial conducted to add evidence to the current European treatment guidelines for adult patients with phenylketonuria.

DETAILED DESCRIPTION:
Phenylketonuria (PKU) is a rare autosomal recessive disorder caused by deficiency of the phenylalanine hydroxylase enzyme leading to an impaired conversion of the amino acid phenylalanine (Phe) to tyrosine. Increased Phe concentrations in blood and brain during childhood can lead to severe intellectual disability, epilepsy and behavioral problems. However, since the introduction of newborn screening and early treatment with a dietary restriction of Phe (low protein diet) and Phe-free protein substitutes (amino acid mixtures) initiated soon after birth, patient with PKU no longer develop profound and irreversible intellectual disability. While there is a wide agreement on the treatment strategy and target Phe concentrations in childhood, no consensus on the safe Phe concentrations in adulthood has been reached so far. Traditionally, the low protein diet had been enforced only during childhood and adolescence, leaving adult patients with PKU "off-diet". Over the last decade, observational and cross-sectional studies associated high Phe in early-treated adult patients with cognitive problems, psychiatric symptoms and behavioral abnormalities. These association studies and one small interventional study led to substantially differing recommendations of national and international guidelines with regard to Phe target levels in adult patients with PKU. One of these guidelines is the highly controversial grade D recommendation of the most recent European guidelines to keep Phe concentrations below 600 μmol/L throughout adulthood. Consequently, the recommendations are not only unequally accepted by the treating metabolic specialists, more than 50 % of adults with PKU exhibit substantial difficulty in maintaining the compliance necessary to reach the recommended target Phe concentrations. Therefore, prospective intervention studies in adult patients with PKU are strongly needed to evaluate the effects of dietary restrictions on cognition, cerebral markers and quality of life. The PICO-Study aims at adding evidence to current guidelines and improving treatment recommendations. To this end, adult patients with PKU will participate in a randomized, placebo-controlled, double-blind, crossover, non-inferiority trial. With the intervention, the project evaluates the impact of temporarily elevated blood Phe levels on cognition and functional properties of the brain of adult patients. Results of the PICO-Study will help to increase knowledge about impaired cognitive functioning and neural abnormalities in adult patients with PKU and will improve guidelines on dietary treatment in these patients. Such guidelines can greatly influence clinical routine as well as patients' adherence to their diet and ultimately their quality of life.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* PKU diagnosed after a positive newborn screening
* Treatment with Phe-restricted diet starting within the first 30 days of life
* Age ≥18 years
* Capable of following the study design
* Written informed consent

Exclusion Criteria:

* Patients with PKU not following a Phe-restricted diet within 6 months before the study
* Phe concentration above 1600 µmol/L within 6 months before the study
* Concomitant disease states suspected to significantly affect primary or secondary outcomes, e. g. untreated vitamin B12 deficiency
* Known or suspected non-compliance, drug or alcohol abuse
* Change in medications likely to significantly interfere with cognitive function testing
* Known or suspected hypersensitivity or allergy to one of the ingredients of the placebo
* Women who are pregnant or intent to get pregnant during the course of the study or who are breast feeding
* Female participants of childbearing potential, not using and not willing to continue using one (or more) highly efficient (Pearl index less than 1) method of contraception for the entire study duration.
* Inability to follow the procedures of the study, e. g. due to language problems (lack of fluency in German or French), psychological disorders, dementia, etc. of the participant.
* Participation in another interventional study within the 30 days preceding and during the present study.
* Previous enrolment into the current study
* Conditions interfering with MRI such as magnetic (metallic) particles in the skull or brain, cardiac pacemaker, deep brain stimulators, cochlear implant, braces or permanent retainers

HEALTHY CONTROLS

Inclusion Criteria:

* Age ≥18 years
* Comparable to patients with regard to age, gender and educational level
* Capable of following the study design
* Written informed consent

Exclusion Criteria:

* Known or suspected drug or alcohol abuse
* Change in medications likely to significantly interfere with cognitive function testing
* Women who are pregnant or intent to get pregnant during the course of the study or who are breast feeding
* Inability to follow the procedures of the study, e. g. due to language problems (lack of fluency in German or French), psychological disorders, dementia, etc. of the participant.
* Participation in another interventional study within the 30 days preceding and during the present study.
* Previous enrolment into the current study
* Conditions interfering with MRI such as magnetic (metallic) particles in the skull or brain, cardiac pacemaker, deep brain stimulators, cochlear implant, braces or permanent retainers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Working memory (accuracy) | After intervention phase 1 (after 4 weeks from baseline)
  Influence of 4 weeks of oral Phe administration vs. Placebo on working memory performance, assessed using accuracy in the n-back task of the Test of Attentional Performance (TAP) in adult patients with phenylketonuria (PKU).
Working memory (accuracy) | After intervention phase 2 (after 12 weeks from baseline)
  Influence of 4 weeks of oral Phe administration vs. Placebo on working memory performance, assessed using accuracy in the n-back task of the Test of Attentional Performance (TAP) in adult patients with PKU.

SECONDARY OUTCOMES:
Working memory (reaction time) | 4 times: baseline, after intervention phase 1 (4 weeks from baseline), after washout (8 weeks from baseline), after intervention phase 2 (12 weeks from baseline)
  Influence of 4 weeks of oral Phe administration vs. Placebo on working memory performance, assessed using reaction time in the n-back task of the Test of Attentional Performance (TAP) in adult patients with PKU.
Inhibition | 4 times: baseline, after intervention phase 1 (4 weeks from baseline), after washout (8 weeks from baseline), after intervention phase 2 (12 weeks from baseline)
  Influence of 4 weeks of oral Phe administration vs. Placebo on inhibition assessed using the third condition of the color-word interference test of the Delis-Kaplan Executive Function System (D-KEFS) in adult patients with PKU.
Cognitive flexibility | 4 times: baseline, after intervention phase 1 (4 weeks from baseline), after washout (8 weeks from baseline), after intervention phase 2 (12 weeks from baseline)
  Influence of 4 weeks of oral Phe administration vs. Placebo on cognitive flexibility assessed using the fourth condition of the color-word interference test of the D-KEFS in adult patients with PKU.
Functional Magnetic Resonance Imaging (fMRI) (working memory) | 4 times: baseline, after intervention phase 1 (4 weeks from baseline), after washout (8 weeks from baseline), after intervention phase 2 (12 weeks from baseline)
  Influence of 4 weeks of oral Phe administration vs. Placebo on intensity of cerebral activation during a working memory task assessed using an n-back task in the MR scanner in adult patients with PKU.
Resting-state fMRI | 4 times: baseline, after intervention phase 1 (4 weeks from baseline), after washout (8 weeks from baseline), after intervention phase 2 (12 weeks from baseline)
  Influence of 4 weeks of oral Phe administration vs. Placebo on strength of functional connectivity in brain regions related to working memory as assessed by resting-state fMRI in adult patients with PKU.
Magnetic Resonance Spectroscopy (MRS) | 4 times: baseline, after intervention phase 1 (4 weeks from baseline), after washout (8 weeks from baseline), after intervention phase 2 (12 weeks from baseline)
  Influence of 4 weeks of oral Phe administration vs. Placebo on brain Phe concentrations as measured by MRS in adult patients with PKU.

OTHER OUTCOMES:
Diffusion Tensor Imaging (DTI) | 4 times: baseline, after intervention phase 1 (4 weeks from baseline), after washout (8 weeks from baseline), after intervention phase 2 (12 weeks from baseline)
  Influence of 4 weeks of oral Phe administration vs. Placebo on white matter integrity assessed using DTI in adult patients with PKU.
Arterial Spin Labeling (ASL) | 4 times: baseline, after intervention phase 1 (4 weeks from baseline), after washout (8 weeks from baseline), after intervention phase 2 (12 weeks from baseline)
  Influence of 4 weeks of oral Phe administration vs. Placebo on cerebral blood flow assessed using ASL in adult patients with PKU.
Structural MRI (cortical thickness) & working memory | Baseline
  Relationship between cortical thickness and working memory (n-back task of the Test of Attentional Performance (TAP)) in adult patients with PKU.
Structural MRI (cortical surface area) & working memory | Baseline
  Relationship between cortical surface area and working memory (n-back task of the Test of Attentional Performance (TAP)) in adult patients with PKU.
Structural MRI (cortical volume) & working memory | Baseline
  Relationship between cortical volume and working memory (n-back task of the Test of Attentional Performance (TAP)) in adult patients with PKU.
Structural MRI (cortical curvature) & working memory | Baseline
  Relationship between cortical curvature and working memory (n-back task of the Test of Attentional Performance (TAP)) in adult patients with PKU.
MRS & working memory | Baseline
  Relationship between brain concentrations of Phe (MRS) and working memory (n-back task of the Test of Attentional Performance (TAP)) in adult patients with PKU.
Blood concentration of Phe & working memory | Baseline
  Relationship between blood concentrations of Phe and working memory (n-back task of the Test of Attentional Performance (TAP)) in adult patients with PKU.
Working memory (accuracy): Patients vs. Controls | Baseline
  Differences in working memory performance, assessed using accuracy in the n-back task of the Test of Attentional Performance (TAP) between adult patients with PKU and healthy controls.
Working memory (reaction time): Patients vs. Controls | Baseline
  Differences in working memory performance, assessed using reaction time in the n-back task of the Test of Attentional Performance (TAP) between adult patients with PKU and healthy controls.
Inhibition: Patients vs. Controls | Baseline
  Differences in inhibition assessed using the third condition of the color-word interference test of the Delis-Kaplan Executive Function System (D-KEFS) between adult patients with PKU and healthy controls.
Cognitive flexibility: Patients vs. Controls | Baseline
  Differences in cognitive flexibility assessed using the fourth condition of the color-word interference test of the D-KEFS between adult patients with PKU and healthy controls.
DTI: Patients vs. Controls | Baseline
  Differences in white matter integrity (DTI) between adult patients with PKU and healthy controls.
fMRI of working memory: Patients vs. Controls | Baseline
  Differences in intensity of cerebral activation during a working memory task assessed using an n-back task in the MR scanner between adult patients with PKU and healthy controls.
ASL: Patients vs. Controls | Baseline
  Differences in cerebral blood flow assessed using ASL between adult patients with PKU and healthy controls.
Resting-state fMRI: Patients vs. Controls | Baseline
  Differences in strength of functional connectivity in brain regions related to working memory as assessed by resting-state fMRI between adult patients with PKU and healthy controls.
Structural MRI (cortical thickness): Patients vs. Controls | Baseline
  Differences in cortical thickness between adult patients with PKU and healthy controls.
Structural MRI (cortical surface area): Patients vs. Controls | Baseline
  Differences in cortical surface area between adult patients with PKU and healthy controls.
Structural MRI (cortical volume): Patients vs. Controls | Baseline
  Differences in cortical volume between adult patients with PKU and healthy controls.
Structural MRI (cortical curvature): Patients vs. Controls | Baseline
  Differences in cortical curvature between adult patients with PKU and healthy controls.
Mood (POMS) | 4 times: baseline, after intervention phase 1 (4 weeks from baseline), after washout (8 weeks from baseline), after intervention phase 2 (12 weeks from baseline)
  Influence of 4 weeks of oral Phe administration vs. Placebo on mood assessed using the short form of the Profile of Mood States (POMS) in adult patients with PKU.
Mood (BDI-II) | 4 times: baseline, after intervention phase 1 (4 weeks from baseline), after washout (8 weeks from baseline), after intervention phase 2 (12 weeks from baseline)
  Influence of 4 weeks of oral Phe administration vs. Placebo on mood assessed using Beck's Depression Inventory (BDI-II) in adult patients with PKU. The total score indicates severity, ranging from 0 (no depression) to 63 (severe depression).
PKU Quality of Life | 4 times: baseline, after intervention phase 1 (4 weeks from baseline), after washout (8 weeks from baseline), after intervention phase 2 (12 weeks from baseline)
  Influence of 4 weeks of oral Phe administration vs. Placebo on the total score in the questionnaire PKU quality of life (PKUQOL) in adult patients with PKU.

CONTACTS AND LOCATIONS:
Overall Officials: Regula Everts, Prof. Dr. phil., Principal Investigator — Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism (UDEM), Inselspital, Bern University Hospital
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism (UDEM), Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trepp R, Muri R, Maissen-Abgottspon S, Haynes AG, Hochuli M, Everts R. Cognition after a 4-week high phenylalanine intake in adults with phenylketonuria - a randomized controlled trial. Am J Clin Nutr. 2024 Apr;119(4):908-916. doi: 10.1016/j.ajcnut.2023.11.007. Epub 2024 Feb 9. PMID 38569786
- [Derived] Trepp R, Muri R, Abgottspon S, Bosanska L, Hochuli M, Slotboom J, Rummel C, Kreis R, Everts R. Impact of phenylalanine on cognitive, cerebral, and neurometabolic parameters in adult patients with phenylketonuria (the PICO study): a randomized, placebo-controlled, crossover, noninferiority trial. Trials. 2020 Feb 13;21(1):178. doi: 10.1186/s13063-019-4022-z. PMID 32054509